CLINICAL TRIAL: NCT04417699
Title: SHORT: SHOrt Course Radiation and TASOX (TAS102 Plus Oxaliplatin) Chemotherapy in Operable Rectal Cancer, a Phase II Trial
Brief Title: SHOrt Course Radiation and TASOX (TAS102 Plus Oxaliplatin) Chemotherapy in Operable Rectal Cancer
Acronym: SHORT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Providence Health & Services (Other)
Collaborators: Taiho Oncology (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021000326
Record Dates: First submitted 2020-05-15; First posted 2020-06-05 (Actual); Results first posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Rectal Cancer
Keywords: SHORT; short course radiation,; TASOX
MeSH Terms: conditions — Rectal Neoplasms | interventions — trifluridine tipiracil drug combination; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- TAS102 plus Oxaliplatin (Experimental): Oxaliplatin 85mg/m2 IV over 2 hours and TAS-102 (35 mg/m2/dose) orally BID
  Interventions: Drug: TAS 102; Drug: Oxaliplatin

INTERVENTIONS:
Drug: TAS 102 — Oral medication over Days 1-5
  Other Names: Tipiracil hydrochloride
Drug: Oxaliplatin — Administered by intravenous infusion over 2 hours on day 1
  Other Names: Eloxatin

SUMMARY:
TASOX can be safely and efficaciously delivered after short course radiation, resulting in significant pathologic downstaging, allowing for an R0 pelvic resection, and providing local control in appropriately selected stage II/III rectal cancer patients treated with contemporary TME-based surgery.

DETAILED DESCRIPTION:
In this phase II study patients will be treated with short-course preoperative irradiation (25 Gy in five fractions of 5 Gy) followed by 6 (six) 2-week cycles of TASOX followed by total mesorectal excision (TME) for patients with resectable rectal cancer (clinical T3c/dN0, T3c/dN1, T2N1). Eligible study subjects include adults who are candidates for curative intent sphincter-sparing surgery and lack high risk features such as tumor encroaching upon the mesorectal-fascia or low tumors who need an Abdominal-Perineal Resection (APR).

ELIGIBILITY:
Inclusion Criteria:

1. Age of at least 18 years.
2. Newly diagnosis of rectal adenocarcinoma.
3. ECOG Performance Status (PS): 0, 1 or 2.
4. Candidate for sphincter-sparing surgical resection prior to initiation of neoadjuvant therapy according to the primary surgeon.
5. Clinical Stage: T1/N1, T2/N1, T3/N1, T3c/dN0.
6. Absence of metastatic disease. Clinical staging is based on physical exam by the primary surgeon, CT scan of the chest/abdomen, and pelvic MRI.

   Node positivity determination: Entry criteria nodes will be measured in short-axis diameter and for the purposes of study entry will be considered positive if 8 mm or greater in short axis.

   Radiographic N2 status is estimated as: 4 or more nodes that measure 8mm or more in short-axis.

   Radiographic N1 status is estimated as: fewer than 4 lymph nodes that measure 8 mm or greater in short axis but 1 or more lymph nodes that measure 8 mm or greater.

   Nodal Metastatic Disease: nodal stations considered suspicious for metastatic disease (M1) for rectal cancer are common iliac, external iliac and inguinal nodes.
7. No evidence of tumor that is adherent to the mesorectal fascia and the ability to perform a curative intent sphincter-sparing TME resection at diagnosis. See exclusion criterion 4
8. The following laboratory values obtained ≤ 28 days prior to registration.

   * Platelet count ≥ 100,000/mm^3
   * Hemoglobin > 8.0 g/dL
   * Total bilirubin ≤ 1.5 x upper limit of normal (ULN)
   * SGOT (AST) ≤ 3 x ULN
   * SGPT (ALT) ≤ 3 x ULN
   * Creatinine ≤1.5 x ULN
9. Negative pregnancy test done ≤ 7 days prior to registration, for women of childbearing potential only.
10. A patient of child-bearing potential is willing to employ adequate contraception. It includes any of the followings: abstinence, oral contraceptives, implantable hormonal contraceptives, or double barrier method (diaphragm plus condom). See exclusion criterion 8
11. Provide informed written consent.
12. Willing to return to enrolling medical site for all study assessments.

Exclusion Criteria:

1. Clinical T4 tumors.
2. Clinical N2 disease estimated as four or more lymph nodes that are ≥8 mm.
3. Primary surgeon indicates need for abdominoperineal (APR) at baseline.
4. Evidence that the tumor is adherent to or invading the mesorectal fascia on imaging studies such that the surgeon would not be able to perform an R0 resection (one with negative margins).

   Distance of the Tumor from the Mesorectal Fascia:

   Patients with tumors with a distance of 1mm or less from the mesorectal fascia reflection have threatened radial margins and are ineligible.
5. Tumor is causing symptomatic bowel obstruction or patients who have had a temporary diverting ostomy are ineligible.
6. Chemotherapy within 5 years prior to registration. (Hormonal therapy is allowable if the disease free interval is ≥ 5 years.)
7. Any prior pelvic radiation.
8. Any of the following because this study involves an agent that has known genotoxic, mutagenic and teratogenic effects:

   * Pregnant women
   * Nursing women
   * Men or women of childbearing potential who are unwilling to employ adequate contraception
9. Co-morbid illnesses or other concurrent disease which, in the judgment of the treating investigator obtaining informed consent, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2022-07-05 (Actual); Primary Completion 2023-12-14 (Actual); Study Completion 2024-02-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hagen Kennecke, MD, Principal Investigator — Providence Health & Services
Locations (4):
- United States (4):
  - University of California, Irvine, Orange, California
  - Columbia University Irving Medical Center/NYPH, New York, New York
  - Providence Portland Medical Center, Portland, Oregon
  - Virginia Mason Medical Center, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TAS102 Plus Oxaliplatin
Started | 13
Completed | 13
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | TAS102 Plus Oxaliplatin
Number analyzed (Participants) | 13
Age, Continuous [Median (Full Range); unit: years] | 66 [43 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 13
Baseline radiologic T stage [Count of Participants; unit: Participants] — Participants in the study were staged and graded based on their clinical and pathological tumor stages, as well as their pathological nodal stages.
  Derivation of the Neoadjuvant response (NAR) score required pathologic staging information from the Total Mesorectal Excision (TME) resection specimen.
  Primary tumor (T): T1, T2, T3, T4: Refers to the size and/or extent of the main tumor. The higher the number after the T, the larger the tumor or the more it has grown into nearby tissues. T's may be further divided to provide more detail, such as T3a and T3b.
  Participants
    cT1 | 0
    cT2 | 0
    cT3a/b | 12
    cT3c/d | 1
    cT4 | 0
Baseline radiologic N stage [Count of Participants; unit: Participants] — Participants in the study were staged and graded based on their clinical and pathological tumor stages and their pathological nodal stages. Derivation of the Neoadjuvant response (NAR) score required pathologic staging information from the TME resection specimen.
  Regional lymph nodes (N): NX: Cancer in nearby lymph nodes cannot be measured; N0: There is no cancer in nearby lymph nodes; N1, N2, N3: Refers to the number and location of lymph nodes that contain cancer. The higher the number after the N, the more lymph nodes that contain cancer.
  Participants
    cN0 | 5
    cN1 | 8
    cN2 | 0
Baseline radiographic M stage [Count of Participants; unit: Participants] — Participants in the study were staged and graded based on their clinical and pathological tumor stages and their pathological nodal stages. Derivation of the Neoadjuvant response (NAR) score required pathologic staging information from the TME resection specimen.
  Distant metastasis (M): MX: Metastasis cannot be measured; M0: Cancer has not spread to other parts of the body; M1: Cancer has spread to other parts of the body.
  Participants
    cM0 | 13
    cM1 | 0

OUTCOME MEASURES:

1. Primary Outcome: Neoadjuvant Response (NAR) Score
Description: Determine whether pre-operative short-course radiation therapy (SRT) and 6 cycles of TASOX offers condensed radiation and total neoadjuvant therapy for intermediate risk rectal cancer. Measurement of efficacy is the NAR score, where the required elements of the NAR score are: clinical tumor stage (cT), pathologic tumor stage (pT), pathological nodal stage (pN).
  For patients with a cCR who opted for non-operative management, for the purposes of the NAR score, those patients were assigned a pT0 and pN0 score if they did not experience tumor regrowth or require subsequent TME surgical resection during the time of the study.
  The NAR score ranges from 0-100, where lower NAR scores are considered favorable as opposed to higher scores which would indicate a worse prognosis.
  NAR calculation as follows:
  NAR=[5 pN- 3(cT-pT)+12]^2/9.61
Time Frame: Through study completion, an average of 6 months
Measure: Mean (Standard Deviation); unit: Calculated score
Arm/Group | TAS102 Plus Oxaliplatin
Number analyzed (Participants) | 13
Calculated score | 9.31 (13.41)

2. Secondary Outcome: Safety and Tolerability
Description: The secondary objective is to describe Incidence of Treatment-Emergent Adverse Events and surgery complications among treated subjects.
Time Frame: Through study completion, an average of 6 months
Measure: Number; unit: participants
Arm/Group | TAS102 Plus Oxaliplatin
Number analyzed (Participants) | 13
participants
  Number of patients who experienced Grade 3 or 4 adverse events | 7
  Number of patients who experienced post-operative complications | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of consent through study completion, an average of 6 months.
Arm/Group | TAS102 Plus Oxaliplatin
All-Cause Mortality (participants affected / at risk) | 1/13
Serious Adverse Events (participants affected / at risk) | 1/13
Other Adverse Events (participants affected / at risk) | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TAS102 Plus Oxaliplatin (N=13)
Diarrhea (Gastrointestinal disorders) | 1 (1) — Bloody diarrhea, required hospitalization.
Rectal Perforation (Gastrointestinal disorders) | 1 (1) — Required hospitalization and treatment delay.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TAS102 Plus Oxaliplatin (N=13)
Abdominal Cramping (Gastrointestinal disorders) | 1 (1)
Abdominal Pain/Discomfort (Gastrointestinal disorders) | 4 (4)
Anosmia (Nervous system disorders) | 1 (1)
Alanine aminotransferase increase (Investigations) | 2 (4)
Aspartate aminotransferase increase (Investigations) | 2 (3)
Blurred vision (Eye disorders) | 1 (1)
Cold sensitivity (General disorders) | 6 (7)
Constipation (Gastrointestinal disorders) | 6 (8)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 9 (12)
Dizziness (Nervous system disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Elevated liver fuction tests (Investigations) | 1 (1)
Fatigue (General disorders) | 6 (7)
Fecal urgency (Gastrointestinal disorders) | 1 (1)
Hypertenson (Vascular disorders) | 1 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Injection site reaction (pain) (General disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Intermittent headaches (Nervous system disorders) | 2 (2)
Joint pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Left flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Leg cramp (Musculoskeletal and connective tissue disorders) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1)
Malaise (General disorders) | 1 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Muscle cramps (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 8 (9)
Neuropathy (Nervous system disorders) | 8 (9)
Neutropenia (Blood and lymphatic system disorders) | 3 (5)
Neutrophil count decreased (Investigations) | 1 (3)
Numbness (Nervous system disorders) | 1 (1)
Discharge on rectum (Gastrointestinal disorders) | 1 (1)
Platelet count decreased (Investigations) | 1 (2)
Radiation cystitis (Gastrointestinal disorders) | 1 (1)
Rectal incontinence (Gastrointestinal disorders) | 1 (2)
Shooting pain in foot (Musculoskeletal and connective tissue disorders) | 1 (1)
Pruritis (Skin and subcutaneous tissue disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Diverticulitis (Gastrointestinal disorders) | 1 (1)
Tachycardia (Vascular disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2)
Thrombophlebitis (Vascular disorders) | 1 (1)
Tingling sensation in fingers (Nervous system disorders) | 1 (1)
Oral dysesthesia (Gastrointestinal disorders) | 1 (1)
Urgency with bowel movements (Gastrointestinal disorders) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1)
Urinary Urgency (Renal and urinary disorders) | 1 (1)
Viral Upper Respiratory Illness (Infections and infestations) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (4)
Weight loss (Investigations) | 1 (1)
White blood cell decreased (Investigations) | 2 (2)
Worsened Anxiety (Psychiatric disorders) | 1 (1)
Worsening GERD (Gastrointestinal disorders) | 1 (1)
Thromboytopenia (Blood and lymphatic system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-06-20): https://cdn.clinicaltrials.gov/large-docs/99/NCT04417699/Prot_SAP_000.pdf